CLINICAL TRIAL: NCT02820298
Title: A Phase 1, Open-label, Randomized, Two-period, Two-treatment, Crossover Study to Evaluate the Effect of A High-Fat Meal on the Pharmacokinetics of Bexagliflozin in Healthy Subjects
Brief Title: Study to Evaluate the Effects of a High-Fat Meal on Bexagliflozin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-481
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Bexagliflozin dosed in fed state, then in fasted state (Experimental): Group 1 subjects will take one dose of 20 mg of bexagliflozin with food on day 1 after an overnight fast and will take a second dose of bexagliflozin without food on day 8 after an overnight fast.
  Interventions: Drug: Bexagliflozin
- Group 2 - Bexagliflozin in fasted state, then in fed state (Experimental): Group 2 subjects will take one dose of 20 mg bexagliflozin without food on day 1 after an overnight fast and will take a second dose of bexagliflozin with food on day 8 after an overnight fast.
  Interventions: Drug: Bexagliflozin

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin tablet, 20 mg
  Other Names: EGT0001442, EGT0001474

SUMMARY:
The purpose of this study was to investigate the effect of a high-fat meal on the levels of bexagliflozin in the blood in healthy subjects.

DETAILED DESCRIPTION:
This was a single center, Phase 1, open-label, 2 × 2 crossover study designed to assess the effects of a high-fat meal on the PK of orally administered bexagliflozin tablets in 18 healthy adults. Subjects were randomized 1:1 to receive bexagliflozin tablets with a high-fat meal on day 1 and without a meal on day 8 after an overnight fast or to receive bexagliflozin tablets without a meal on day 1 after an overnight fast and with a high-fat meal on day 8.

Subjects were admitted to the clinic on the day before dosing in each treatment period, and stayed in the clinic until 48 h post-dose.

The subjects dosed in the fed state received an oral bexagliflozin tablet, 20 mg, 30 min after starting to consume a high-fat meal following an overnight fast. The meal was to be ingested in its entirety over an approximate 25-minute period, such that it was completed at least 5 minutes prior to the scheduled time of bexagliflozin dosing for the fed state treatment. Subjects dosed in the fasting state received an oral bexagliflozin tablet, 20 mg, after an overnight fast.

Blood samples for bexagliflozin plasma concentrations were collected at 0 h (pre-dose), and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose. Urine collection in 12 h batches was performed at pre-dose (-12 to 0 h on day 0 and day 7), and at post-dose (0 to 12 h, 12 to 24 h, 24 to 36 h, and 36 to 48 h) intervals.

ELIGIBILITY:
Each subject had to meet the following criteria to be eligible for the study:

1. Subjects who were between 18-65 years of age with body-mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2.
2. Male subjects who were surgically sterile or male subjects who were not surgically sterile must have agreed to refrain from donating sperm and used appropriate birth control for a period of 30 days after discharge from the clinic.
3. Female subjects of childbearing potential who were willing to use an adequate method of contraception and to not become pregnant for the duration of the study.
4. Female subjects who were surgically sterile or postmenopausal were eligible if they tested negative on the urine pregnancy test.
5. Subjects who were non-smokers for at least 3 months prior to screening.
6. Subjects with adequate venous access at multiple sites in both arms.
7. Subjects who were willing and able to be confined to the clinical research facility as required by the Protocol.
8. Subjects who had the ability to comprehend and willingness to provide written informed consent in accordance with institutional and regulatory guidelines.

Subjects who met any of the following criteria were excluded from the study:

1. Subjects who were determined by the Investigator or sub-Investigator to be unsuitable for participating in the study based on medical conditions.
2. Female subjects who were nursing or pregnant.
3. Subjects with a clinically significant history of allergy to drugs or latex.
4. Subjects with a history of alcohol or drug dependence in the last 12 months.
5. Subjects who had 400 mL of whole blood collected within four months or 200 mL of whole blood collected within one month of the screening test.
6. Subjects who had blood component collection within 14 days prior to the screening test.
7. Subjects who had used prescription or over-the-counter drugs within 14 days prior to the first dose.
8. Subjects who had used vitamin preparations or supplements (including St. John's Wort and ginseng) within 14 days prior to the first dose.
9. Subjects who had undergone strenuous activity within 72 hours prior to Day 1 in each period.
10. Subjects who were unable (e.g., food intolerance) or unwilling to consume a high-fat breakfast within 25 minutes.
11. Subjects who had been treated with an investigational drug within 30 days or 7 half-lives of the investigational drug, whichever was longer, prior to the first dose of study drug in this trial.
12. Subjects who had previously received EGT0001474 or bexagliflozin, or any other SGLT2 inhibitors within 3 months from screening.
13. Subjects whose screening electrocardiogram (ECG) demonstrated any one of the following: heart rate >100 bpm, QRS >120 msec, QTc >470 msec (corrected by Bazett's formula), PR >220 msec (a subject with PR >220 msec would generally be excluded but exceptions may have been allowed at the discretion of the Investigator), or any rhythm that was not sinus rhythm, sinus bradycardia, or sinus arrhythmia.
14. Subjects whose sitting blood pressure was above 140/90 mmHg at screening.
15. Subjects who had a positive result of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, urinary drug or urinary cotinine test.
16. Subjects with known human immunodeficiency virus (HIV) disease.
17. Subjects with abnormal vital signs, laboratory values, symptoms or signs that were deemed clinically significant by the Investigator.
18. Subjects who had had a febrile illness within 5 days prior to the first dose of study medication.
19. Subjects vaccinated within 30 days prior to the first dose of medication.
20. Detectable urine glucose at screening (trace or greater).
21. Subjects with eGFR <90 mL/min/1.73 m2 or a history of kidney transplant.
22. Subjects with digestion problems, including gastroesophageal reflux disease, irritable bowel syndrome, gastroparesis, and any other disorder deemed by the Investigator to be clinically significant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Williams, M.D., Study Director — Davita Clinical Research
Locations (1):
- Denver Clinical Research Unit, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bexagliflozin Administered in Fed Condition, Then in Fasted Condition: Subjects were dosed with bexagliflozin tablet, 20 mg, with a high-fat meal on day 1 and a second dose of bexagliflozin tablet in fasted state on day 8.
- Bexagliflozin Administered in Fasted Condition, Then in Fed Condition: Subjects were dosed with bexagliflozin tablet, 20 mg, in fasted state on day 1 and second dose of bexagliflozin tablet with a high-fat meal on day 8
Period: Overall Study
Arm/Group | Bexagliflozin Administered in Fed Condition, Then in Fasted Condition | Bexagliflozin Administered in Fasted Condition, Then in Fed Condition
Started | 13 | 12
Completed | 12 | 10
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin Administered in Fed Condition, Then in Fasted Condition | Bexagliflozin Administered in Fasted Condition, Then in Fed Condition | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (10.1) | 31.8 (10.6) | 31.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 8 | 9 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 75.05 (14.65) | 71.58 (12.42) | 73.38 (13.46)
Height [Mean (Standard Deviation); unit: cm] | 173.6 (9.3) | 171.1 (8.8) | 172.4 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Plasma Concentration)
Description: Blood samples (2 mL) for bexagliflozin plasma concentrations were collected at 0 h (pre-dose), and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose (days 1-3 in treatment period 1 and days 8-10 in treatment period 2, respectively)
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose
Population: The PK Population included all randomized subjects who received study drug and who had sufficient plasma bexagliflozin measurements to derive at least one PK parameter following dosing.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Bexagliflozin Tablet Dosed in Fed Condition: Subjects were dosed with bexagliflozin tablet, 20 mg, with a high-fat meal on day 1 after an overnight fast and a second dose of bexagliflozin without a high-fat meal on day 8 after an overnight fast.
- Bexagliflozin Tablet Dosed in Fasted Condition: Subjects were dosed with bexagliflozin tablet, 20 mg, without a high-fat meal on day 1 after an overnight fast and a second dose of bexagliflozin with a high-fat meal on day 8 after an overnight fast.
Arm/Group | Bexagliflozin Tablet Dosed in Fed Condition | Bexagliflozin Tablet Dosed in Fasted Condition
Number analyzed (Participants) | 23 | 24
ng/mL | 176.1 (30.6) | 133.7 (42.5)
Statistical Analysis 1: Comparison: Bexagliflozin Tablet Dosed in Fed Condition vs Bexagliflozin Tablet Dosed in Fasted Condition; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 131.41, 90% CI 2-sided [117.03 to 147.56] — Ratio of Geometric LSM is the ratio of exponentiated mean difference of log-transformed PK parameter. Confidence interval from ANOVA (linear mixed-effects model) with treatment, period, and sequence as fixed effects, and subject as a random effect

2. Primary Outcome: Tmax (Time of Maximum Observed Plasma Concentration)
Description: as for outcome 1
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose
Population: PK population
Measure: Median (Full Range); unit: hours
Groups:
- Bexagliflozin Tablet Dosed in Fed Condition: Subjects were dosed with bexagliflozin tablet with a high-fat meal
- Bexagliflozin Tablet Dosed in Fasted Condition: Subjects were dosed with bexagliflozin tablet in fasted condition
Arm/Group | Bexagliflozin Tablet Dosed in Fed Condition | Bexagliflozin Tablet Dosed in Fasted Condition
Number analyzed (Participants) | 23 | 24
hours | 5.0 [3 to 8] | 3.5 [2 to 5]

3. Primary Outcome: AUC0-t (Area Under the Plasma Concentration-time Curve From Time 0 to t)
Description: as for outcome 1
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose
Population: PK population
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Bexagliflozin Tablet Dosed in Fed Condition: Subjects were dosed with bexagliflozin tablet, 20 mg, with a high-fat meal after an overnight fast.
- Bexagliflozin Dosed in Fasted Condition: Subjects were dosed with bexagliflozin tablet, 20 mg, in fasted condition.
Arm/Group | Bexagliflozin Tablet Dosed in Fed Condition | Bexagliflozin Dosed in Fasted Condition
Number analyzed (Participants) | 23 | 24
h*ng/mL | 1222.7 (26.8) | 1074.2 (33.0)
Statistical Analysis 1: Comparison: Bexagliflozin Tablet Dosed in Fed Condition vs Bexagliflozin Dosed in Fasted Condition; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 110.29, 90% CI 2-sided [103.91 to 117.06] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: AUC0-∞ (Area Under the Plasma Concentration-time Curve From Time 0 to ∞)
Description: as for outcome 1
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose
Population: PK population
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Bexagliflozin Tablet Dosed in Fed Condition: Group 1 subjects will take one dose of bexagliflozin tablet, 20 mg, with a high-fat meal on day 1 after an overnight fast and a second dose of bexagliflozin without a high-fat meal on day 8 after an overnight fast.
- Bexagliflozin Dosed in Fasted Condition: Group 2 subjects will take one dose of bexagliflozin tablet, 20 mg, without a high-fat meal on day 1 after an overnight fast and a second dose of bexagliflozin with a high-fat meal on day 8 after an overnight fast.
Arm/Group | Bexagliflozin Tablet Dosed in Fed Condition | Bexagliflozin Dosed in Fasted Condition
Number analyzed (Participants) | 23 | 24
ng*h/mL | 1258.7 (5.8) | 1161.8 (5.7)
Statistical Analysis 1: Comparison: Bexagliflozin Tablet Dosed in Fed Condition vs Bexagliflozin Dosed in Fasted Condition; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 108.34, 90% CI 2-sided [102.48 to 114.54] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: T1/2 (Apparent Terminal Elimination Half-life)
Description: Whole venous blood samples of 3 mL were collected from a peripheral vein prior to dosing and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h after administration of bexagliflozin; On Day 1 and Day 5 for Study 1, Day 1 and Day 6 for Study 2, Day 1 and Day 4 for Study 3. The pharmacokinetic parameters were estimated from the bexagliflozin plasma concentration data for each subject by non-compartmental analysis (NCA).
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Bexagliflozin Tablet Dosed in Fed Condition | Bexagliflozin Dosed in Fasted Condition
Number analyzed (Participants) | 23 | 24
hours | 10.1 (28.2) | 11.7 (38.0)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from Day 0 up to Day 10
Groups:
- Bexagliflozin Tablet Dosed in Fasted Condition: Subjects were dosed with bexagliflozin tablet, 20 mg, in fasted condition after an overnight fast
Arm/Group | Bexagliflozin Tablet Dosed in Fed Condition | Bexagliflozin Tablet Dosed in Fasted Condition
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 5/23 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin Tablet Dosed in Fed Condition (N=23) | Bexagliflozin Tablet Dosed in Fasted Condition (N=24)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal congestion (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has no right to publish the results.

DOCUMENTS (2):
  • Study Protocol (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT02820298/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT02820298/SAP_001.pdf